CLINICAL TRIAL: NCT04246411
Title: Ultrasound-guidance Versus Auscultation to Confirm Optimal Insertion Depth of the Cuffless Oral Ring-Adair-Elwyn (RAE) Endotracheal Tube in Pediatric Patients
Brief Title: Ultrasound vs. Auscultation for Optimal Depth of the Cuffless RAE Tube
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was confirmed that cuffed RAE tubes with small diameter could be used, so there was no reason to use RAE cuffless tubes.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: US-RAE
Record Dates: First submitted 2020-01-14; First posted 2020-01-29 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Intubation Complication; Child; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Active Comparator): Ultrasound-guided detection of endobronchial intubation depth by loss of lung sliding sign in the left lung field
  Interventions: Behavioral: Ultrasound-guided determination of cuffless RAE tube depth
- Auscultation (Placebo Comparator): Auscultation-guided detection of endobronchial intubation depth by loss of breathing sound in the left lung field
  Interventions: Behavioral: Auscultation-guided determination of cuffless RAE tube depth

INTERVENTIONS:
Behavioral: Ultrasound-guided determination of cuffless RAE tube depth — 1. Measurement of "Carina-T2 mid-vertebra length" from preoperative Cheat PA
  2. Ultrasound-guided detection of endobronchial intubation depth by loss of lung sliding sign in the left lung field.
  3. Withdrawal of the cuffless RAE tube using the "Carina-T2 mid-vertebra length" for optimal positioning
  Arms: Ultrasound
Behavioral: Auscultation-guided determination of cuffless RAE tube depth — 1. Measurement of "Carina-T2 mid-vertebra length" from preoperative Cheat PA
  2. Auscultation-guided detection of endobronchial intubation depth by loss of breathing sound in the left lung field
  3. Withdrawal of the cuffless RAE tube using the "Carina-T2 mid-vertebra length" for optimal positioning
  Arms: Auscultation

SUMMARY:
The aim of this study is to compare the ultrasound-guidance versus auscultation to confirm optimal insertion depth of the cuffless oral Ring-Adair-Elwyn (RAE) endotracheal tube in pediatric patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children age under 7 years
* Undergoing general anesthesia
* Endobronchial intubation with cuffless oral RAE tube

Exclusion Criteria:

* Pulmonary disease
* Active upper respiratory tract infection
* History of upper or lower respiratory tract infection within 2 weeks
* Emergent operation
* Unstable vital sign

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of optimal location of the cuffless Oral RAE tube (%) | during operation (until endotracheal extubation) up to 18 hour after induction
  The distance between the tip of cuffless RAE tube and right pulmonary artery is within the -5mm ~ +5mm value of the distance between the T2 mid-vertebra and carina (optimal depth)

SECONDARY OUTCOMES:
M-distance (between the carina and the T2 mid-vertebra) | during operation up to 18 hour after induction
  The distance between T2 mid-vertebra and the carina)
Distance between the optimal depth and the relocated depth | during operation up to 18 hour after induction
  Distance between the optimal depth and the relocated depth
Subglottic diameter at the cricoid cartilage level | during operation
  Subglottic diameter at the cricoid cartilage level using neck US
ID and OD of optimal cuffless oral RAE tube | during operation up to 18 hour after induction
  Internal and external diameter of optimal cuffless oral RAE tube
Time from intubation to confirming the tube depth | during operation up to 18 hour after induction
  Time from intubation to confirming the tube depth (seconds)
Distance between the optimal depth and the manufacturer's recommended depth | during operation up to 18 hour after induction
  Distance between the optimal depth and the manufacturer's recommended depth
Airway leakage pressure | during operation up to 18 hour after induction
  Airway leakage pressure measured by manual ventilation with APL(Adjustable pressure-limiting) valve
Incidence of the intraoperative airway-related events | during operation up to 18 hour after induction
  accidental extubation, endobronchial intubation, desaturation (SpO2 < 95%), etc
Incidence of the airway-related symptoms after extubation | up to 18 hour after induction
  hoarseness, stridor, laryngospasm, chest retraction, etc

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD.PhD, Principal Investigator — Professor, Seoul National University Hospital
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altun D, Orhan-Sungur M, Ali A, Ozkan-Seyhan T, Sivrikoz N, Camci E. The role of ultrasound in appropriate endotracheal tube size selection in pediatric patients. Paediatr Anaesth. 2017 Oct;27(10):1015-1020. doi: 10.1111/pan.13220. Epub 2017 Aug 28. PMID 28846176
- [Background] Ahn JH, Kwon E, Lee SY, Hahm TS, Jeong JS. Ultrasound-guided lung sliding sign to confirm optimal depth of tracheal tube insertion in young children. Br J Anaesth. 2019 Sep;123(3):309-315. doi: 10.1016/j.bja.2019.03.020. Epub 2019 Apr 12. PMID 30987765